CLINICAL TRIAL: NCT03135015
Title: Acute Effect of HP-211 (Axulin) on Blood Glucose and Serum Insulin Responses in Healthy Lean and Overweight Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Housey Healthcare ULC (Industry)
Collaborators: Glycemic Index Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIL-1665
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Results first posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-01

CONDITIONS: Insulin Resistance, Diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Each participant in 2 participant groups will undergo each of 6 treatments
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Capsule treatments will be fully blinded. Tablet treatments will be open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lean Participants (Other): Participants with BMI >18.5 and <25.0kg/m²
  Interventions: Other: Placebo capsules; Other: 2g capsules; Other: 4g capsules; Other: Water Control; Other: 2g tablets; Other: 4g tablets
- Overweight/Obese Participants (Other): Participants with BMI ≥25.0 and <35.0kg/m²
  Interventions: Other: Placebo capsules; Other: 2g capsules; Other: 4g capsules; Other: Water Control; Other: 2g tablets; Other: 4g tablets

INTERVENTIONS:
Other: Placebo capsules — 250ml water with 16 x 250mg placebo capsules
Other: 2g capsules — 250ml water with 8 x 250mg capsules containing Axulin powder plus 8 x 250mg placebo capsules
Other: 4g capsules — 250ml water with 16 x 250mg capsules containing Axulin powder
Other: Water Control — 250ml water
Other: 2g tablets — 250ml water with 2 x 1g tablets containing Axulin powder
Other: 4g tablets — 250ml water with 4 x 1g tablets containing Axulin powder

SUMMARY:
Blood sugar levels are controlled by insulin, a hormone made by cells in the pancreas. After a meal, carbohydrates are broken down into glucose (blood sugar) which is absorbed from the intestine into the blood leading to a rise in glucose which triggers the secretion of insulin. Insulin binds to cells in the liver, muscle and fat, triggering them to take up glucose and bring the blood glucose level back to normal.

A high blood sugar level is known as diabetes. The most common form of diabetes, type 2 diabetes, is caused by insulin resistance; that is, a reduced ability of insulin to stimulate glucose uptake into cells. The body compensates for insulin resistance by making more insulin; type 2 diabetes occurs when the pancreas can no longer make enough insulin to control blood glucose. The high blood glucose and insulin levels lead to long-term complications such as heart attacks, kidney failure, reduced sensation and poor circulation in the feet and legs. Reducing blood glucose levels with oral medications and insulin reduces risk of diabetic complications. There are several types of oral medications available for treating diabetes; however, they do not always control blood glucose adequately. In addition, these drugs have complications and are not used to treat insulin resistance and prediabetes - a condition when blood glucose is higher than normal but not high enough to be classified as diabetes. Prediabetes often progresses to diabetes over a period of months or years. Effective and safe treatments for prediabetes could prevent or delay the onset of diabetes.

Axulin is a natural health product consisting of a mixture of extracts - derived from herbs and vegetables present in normal diets - which has been shown in cell culture and in animal studies to increase the ability of insulin to stimulate glucose uptake into cells. The active ingredient in Axulin is a botanical extract designated HP-211. Thus, HP-211 may reduce the blood glucose and insulin levels of subjects without diabetes after eating. HP-211 may also reduce glucose and insulin responses to a larger extent in insulin-resistant as compared to insulin-sensitive subjects.

Subjects will take 0g, 2g, or 4g of capsules or tablets in the morning after an overnight fast; 40 minutes later they will consume 75g glucose dissolved in 300ml water. Blood glucose, insulin and fats will be measured before and for 2 hours after the glucose drink.

DETAILED DESCRIPTION:
After consumption of a meal, pancreatic secretions of various digestive enzymes results in the breakdown of carbohydrates into monosaccharides including glucose. These sugars are subsequently absorbed through the intestinal lumen, resulting in an increased plasma glucose concentration. In response to high glucose levels, pancreatic beta-cells are stimulated to release the hormone insulin which circulates through the bloodstream and binds to insulin-responsive cells including adipocytes (fat tissue), myocytes (muscle tissue), and hepatocytes (liver). The resulting insulin-mediated signaling cascade initiates intracellular glucose uptake within peripheral tissues leading to a corresponding decrease in circulating plasma glucose.

In insulin responsive cells glucose uptake stimulation begins after the binding of insulin to Insulin Receptors (IR), which are found on the membrane surface of cells in insulin responsive tissues such as fat, muscle and liver. The IR consists of an extracellular domain which binds to insulin, and an intracellular domain that has a protein tyrosine kinase activity. The binding of Insulin to the IR initiates a series of auto-phosphorylation events within the protein kinase domain that permit interaction and phosphorylation of downstream signaling proteins in the cell that mediate the cellular response to insulin. The resulting signaling complex includes proteins in the Insulin Receptor Substrate (IRS) family known as IRS-1 and IRS-2. These key targets of the insulin signaling pathway link IR activation to downstream signaling cascades that mediate intracellular processes including GLUT4-mediated glucose uptake.

Prediabetes and Type II diabetes involve an impaired post-receptor response to insulin that hinders the glucose uptake response after meal consumption. Chronic hyperglycemia and the resulting compensatory hyperinsulinemia promote a cohort of acute and chronic sequelae including cardiovascular disease, liver complications, central nervous system degeneration and hyperglycemic osmotic stress. Axulin is a natural health product consisting of a mixture of extracts from herbs and vegetables present in normal diets which was identified by screening more than 100,000 compounds and extracts in a patented cell-culture based assay system targeting the IRS proteins. In vitro, Axulin's active ingredient, HP-211, has marked effects on the IRS-2 branch of the insulin signaling cascade to enhance downstream insulin signaling. HP-211 has been shown in animal models to increase glucose uptake in peripheral tissues and decrease circulating blood glucose and triglyceride concentrations. Regular supplementation of the diet with Axulin would be expected to reduce the incidence of associated prediabetic and diabetic complications, resulting in an increased quality of life for patients without resorting to current anti-diabetic prescription drugs such as metformin and others that may have substantial unwanted side effects in patients.

HYPOTHESES Axulin will reduce postprandial glucose and insulin responses in a dose-dependent fashion in healthy subjects without diabetes. The reduction in glucose and insulin will be relatively greater in insulin-resistant than insulin-sensitive subjects.

Subjects will take 0g, 2g, or 4g of capsules or tablets in the morning after an overnight fast; 40 minutes later they will consume 75g glucose dissolved in 300ml water. Blood glucose, insulin and triglycerides will be measured fasting and at intervals for 2 hours after the glucose drink.

ELIGIBILITY:
Inclusion Criteria:

* Participants taking stable doses (for at least 4 weeks of signing the consent form) of the birth control pill, thyroxin replacement therapy, statins, fibrates, cholesterol absorption inhibitors, anti-hypertensive medications, asprin, non-steroidal anti-inflammatories and/or mild anxiolytics or sedatives can be included.

Exclusion Criteria:

* Fasting serum glucose >6.9mmol/L (124mg/dL)
* HbA1c >6.4%
* Fasting serum triglycerides >4.5 mmol/L (399 mg/dL)
* Fasting LDL cholesterol >4.99 mmol/L (192 mg/dL)
* Blood pressure >149 systolic or >89 diastolic
* Serum creatinine, or aspartate- or alanine transaminases >1.2 times upper limit of normal
* White cell count, red blood cell count, hemoglobin or hematocrit outside normal range
* Hospitalization for surgery or a medical condition within 3 months of signing the consent form
* Use of any drug to treat diabetes
* Use of medications other than those listed above or the presence of any condition which might, in the opinion of Dr. Wolever, either: 1) make participation dangerous to the subject or to others, or 2) affect the results
* Allergy or sensitivity to tarragon, chromium, escarole, lettuce, microcrystalline cellulose, inulin, food colouring (FD&C Yellow#5 and Blue#1) or vegetable-based capsules (silicon dioxide, titanium dioxide, hydroxypropylmethylcellulose)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — Glycemic Index Laboratories, Inc
Locations (1):
- Glycemic Index Laboratories, Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 26-APRIL-2017 to 24-MAY-2017 at GI Labs (20 Victoria St., Toronto ON, M5C 2N8).
Pre-assignment Details: A screening visit was conducted to ensure each participant met inclusion/exclusion criteria for the study. Participants that qualified for the study were separated into either the lean or the overweight group as per protocol (11 subjects/arm).Participants were assigned to a randomization schedule in order of enrollment within each group.
Groups:
- Lean Participants: Participants with BMI >18.5 and <25.0kg/m². All participants received each of the 6 interventions in a randomized manner.
- Overweight/Obese Participants: Participants with BMI ≥25.0 and <35.0kg/m². All participants received each of the 6 interventions in a randomized manner.
Period: Overall Study
Arm/Group | Lean Participants | Overweight/Obese Participants
Started | 11 | 11
Water Control | 9 | 11
Placebo Capsules | 9 | 11
2g Capsules | 9 | 11
4g Capsules | 9 | 11
2g Tablets | 9 | 11
4g Tablets | 9 | 11
Completed | 9 | 11
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: The analysis of baseline characteristics includes all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lean Participants | Overweight/Obese Participants | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (9.1) | 45 (13) | 39.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 5 | 7 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 2 | 0 | 2
  Caucasian | 4 | 7 | 11
  Korean | 1 | 0 | 1
  Latin American | 1 | 0 | 1
  Chinese | 2 | 1 | 3
  South Asian | 1 | 2 | 3
  South East Asian | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 11 | 11 | 22
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 22.2 (1.7) | 28.5 (2.7) | 25.4 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Area Under The Curve (AUC) for Blood Glucose 0-2 Hours
Description: Percentage change in the incremental area under the glucose response curve (AUC) after 75g glucose for capsules and tablets containing Axulin powder relative to the water control. Incremental AUC is the AUC below the curve above the fasting level; area below fasting is ignored. Percentage change will be calculated as 100 x (A-P)/P where A and P are the mean AUC's after Axulin and water control treatments, respectively. The blinded AUC results for the 6 treatments will be subjected to repeated measures analysis of variance (ANOVA) examining for the main effects of treatment and participant-group, and treatment*group interaction. After demonstration of significant heterogeneity among the 6 coded treatments, differences between individual means will be assessed using Tukey's test to adjust for multiple comparisons. The code will be broken after this analysis has been done. The percentage changes will be considered to be significant if the difference in mean AUC is significant.
Time Frame: 0, 15, 30, 45, 60, 90, and 120 minutes post-dose
Population: The analysis of primary outcome data is based on all randomized subjects who received this intervention and for whom primary outcome data is known. There is no missing value imputation.
Measure: Least Squares Mean (Standard Error); unit: mmol x min/L
Groups:
- Water Control: All Participants randomized to receive 250ml water.
- 2g Capsules: All Participants randomized to receive 250ml water with 8 x 250mg capsules containing Axulin powder plus 8 x 250mg placebo capsules.
- 4g Capsules: All Participants randomized to receive 250ml water with 16 x 250mg capsules containing Axulin powder.
- Placebo Capsules: All Participants randomized to receive 250ml water.with 16 x 250mg placebo capsules.
- 2g Tablets: All Participants randomized to receive 250ml water with 2 x 1g tablets containing Axulin powder.
- 4g Tablets: All Participants randomized to receive 250ml water with 4 x 1g tablets containing Axulin powder.
Arm/Group | Water Control | 2g Capsules | 4g Capsules | Placebo Capsules | 2g Tablets | 4g Tablets
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
mmol x min/L | 301.09 (27.6405) | 258.66 (27.6405) | 248.63 (27.6405) | 274.13 (27.1449) | 325.73 (0.7879) | 306.19 (52.3273)
Statistical Analysis 1: Comparison: Water Control vs 2g Capsules; The blinded AUC results for the 6 treatments will be subjected to repeated measures analysis of variance (ANOVA) examining for the main effects of treatment and participant-group, and treatment*group interaction. After demonstration of significant heterogeneity among the 6 coded treatments, differences between individual means will be assessed using Tukey's test to adjust for multiple comparisons; Test type: Other; p = 0.1146, t-test, 2 sided; Percentage Change from Control = -14.09
Statistical Analysis 2: Comparison: Water Control vs 4g Capsules; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0519, t-test, 2 sided; Percentage Change from Control = -17.42
Statistical Analysis 3: Comparison: Water Control vs Placebo Capsules; [analysis description as in outcome 1, analysis 1]; Test type: Other; Percentage Change from Control = -8.95

2. Secondary Outcome: Blood Glucose Area Under The Curve (AUC) 0-2 Hours
Description: Incremental area under the blood glucose response curve (AUC) is the AUC below the glucose response curve above the fasting level; area below fasting is ignored. The blinded AUC results for the 6 treatments will be subjected to repeated measures analysis of variance (ANOVA) examining for the main effects of treatment and participant-group, and treatment*group interaction. After demonstration of significant heterogeneity among the 6 coded treatments, differences between individual means will be assessed using Tukey's test to adjust for multiple comparisons. The code will be broken after this analysis has been done.
Time Frame: 0, 15, 30, 45, 60, 90, and 120 minutes post-dose
Population: The analysis of secondary outcome data is based on all randomized subjects who received this intervention and for whom secondary outcome data is known. There is no missing value imputation.
Measure: Least Squares Mean (Standard Error); unit: mmol x min/L
Groups:
- 2g Capsules: All Participants randomized to receive 250ml water.with 8 x 250mg capsules containing Axulin powder plus 8 x 250mg placebo capsules.
Arm/Group | Water Control | 2g Capsules | 4g Capsules | Placebo Capsules | 2g Tablets | 4g Tablets
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
mmol x min/L | 301.09 (27.6405) | 258.66 (27.6405) | 248.63 (27.6405) | 274.13 (27.1449) | 325.73 (0.7879) | 306.19 (52.3273)
Statistical Analysis 1: Comparison: Water Control vs 2g Capsules; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.1146, t-test, 2 sided
Statistical Analysis 2: Comparison: Water Control vs 4g Capsules; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0519, t-test, 2 sided

3. Secondary Outcome: Serum Insulin Area Under The Curve (AUC) 0-2 Hours
Description: Incremental area under the serum insulin response curve (AUC) is the AUC below the insulin response curve above the fasting level; area below fasting is ignored. The blinded AUC results for the 6 treatments will be subjected to repeated measures analysis of variance (ANOVA) examining for the main effects of treatment and participant-group, and treatment*group interaction. After demonstration of significant heterogeneity among the 6 coded treatments, differences between individual means will be assessed using Tukey's test to adjust for multiple comparisons. The code will be broken after this analysis has been done.
Time Frame: 0, 15, 30, 45, 60, 90, and 120 minutes post-dose
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: uU x min/ml
Arm/Group | Water Control | 2g Capsules | 4g Capsules | Placebo Capsules | 2g Tablets | 4g Tablets
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
uU x min/ml | 4379.31 (625.35) | 4005.61 (634.61) | 4787.44 (634.61) | 4135.18 (493.30) | 4452.09 (461.79) | 4381.71 (545.47)
Statistical Analysis 1: Comparison: Water Control vs 2g Capsules; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.5827, t-test, 2 sided
Statistical Analysis 2: Comparison: Water Control vs 4g Capsules; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.5485, t-test, 2 sided

4. Secondary Outcome: Percentage Change in Area Under The Curve (AUC) for Serum Insulin 0-2 Hours
Description: Percentage change in the incremental area under the insulin response curve (AUC) after 75g glucose for the capsules containing Axulin powder relative to the water control. Incremental AUC is the AUC below the curve above the fasting level; area below fasting is ignored. Percentage change will be calculated as 100 x (A-P)/P where A and P are the mean AUC's after Axulin and water control treatments, respectively. The blinded AUC results for the 6 treatments will be subjected to repeated measures analysis of variance (ANOVA) examining for the main effects of treatment and participant-group, and treatment*group interaction. After demonstration of significant heterogeneity among the 6 coded treatments, differences between individual means will be assessed using Tukey's test to adjust for multiple comparisons. The code will be broken after this analysis has been done. The percentage changes will be considered to be significant if the difference in mean AUC is significant.
Time Frame: 0, 15, 30, 45, 60, 90, and 120 minutes post-dose
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: uU x min/ml
Arm/Group | Water Control | 2g Capsules | 4g Capsules | Placebo Capsules | 2g Tablets | 4g Tablets
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
uU x min/ml | 4379.31 (625.35) | 4005.61 (634.61) | 4787.44 (634.61) | 4135.18 (493.30) | 4452.09 (461.79) | 4381.71 (545.47)
Statistical Analysis 1: Comparison: Water Control vs 2g Capsules; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.5827, t-test, 2 sided; Percentage Change from Control = -8.53
Statistical Analysis 2: Comparison: Water Control vs 4g Capsules; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.5485, t-test, 2 sided; Percentage Change from Control = 9.32

5. Secondary Outcome: Insulinogenic Index
Description: Insulinogenic Index is an index of the ability of a change in blood glucose to stimulate an increase in serum insulin. It is a unitless measure with higher numbers indicating improved beta cell function. It is calculated by dividing the change in serum insulin between 0 and 30 minutes by the change in blood glucose between 0 and 30 minutes.
Time Frame: Baseline and 30 minutes
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Insulinogenic Index
Arm/Group | Water Control | 2g Capsules | 4g Capsules | Placebo Capsules | 2g Tablets | 4g Tablets
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Insulinogenic Index | 11.462 (2.276) | 15.540 (2.769) | 17.436 (2.879) | 15.059 (3.401) | 13.785 (2.772) | 13.580 (2.586)
Statistical Analysis 1: Comparison: Water Control vs 2g Capsules; Test type: Other; p = 0.1234, t-test, 2 sided
Statistical Analysis 2: Comparison: Water Control vs 4g Capsules; Test type: Other; p = 0.0331, t-test, 2 sided

6. Secondary Outcome: Matsuda Insulin Sensitivity Index
Description: Matsuda Insulin Sensitivity Index is an index of whole body insulin sensitivity derived from glucose and insulin responses after a 75g Oral Glucose Tolerance Test (OGTT). It is calculated by 10000 divided by the square root of (FG*FI*MG*MI) where FG is fasting glucose, FI is fasting insulin, MG is the mean AUC for blood glucose at 0, 30, 60, 90 and 120 minutes and MI is the mean AUC for serum insulin at 0, 30, 60, 90 and 120 minutes.
Time Frame: 0, 30, 60, 90, and 120 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Matsuda Insulin Sensitivity Index
Arm/Group | Water Control | 2g Capsules | 4g Capsules | Placebo Capsules | 2g Tablets | 4g Tablets
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Matsuda Insulin Sensitivity Index | 206.116 (25.116) | 165.289 (20.926) | 155.64 (15.775) | 186.468 (23.788) | 167.004 (15.441) | 189.457 (17.999)
Statistical Analysis 1: Comparison: Water Control vs 2g Capsules; Test type: Other; p < 0.0500, t-test, 2 sided
Statistical Analysis 2: Comparison: Water Control vs 4g Capsules; Test type: Other; p = 0.0568, t-test, 2 sided

7. Secondary Outcome: ISSI-2 Index of Beta-cell Function
Description: Insulin Secretion-Sensitivity Index-2 (ISSI-2) is an index of β-cell function with insulin secretion adjusted for whole body insulin sensitivity. It is calculated by the total area under the curve for serum insulin divided by the area under the curve for blood glucose, and that result times the Matsuda insulin sensitivity index (defined above).
Time Frame: 0, 30, 60, 90, and 120 minutes post-dose
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Insulin Secretion-Sensitivity Index-2
Arm/Group | Water Control | 2g Capsules | 4g Capsules | Placebo Capsules | 2g Tablets | 4g Tablets
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Insulin Secretion-Sensitivity Index-2 | 816.475 (50.412) | 705.232 (49.158) | 773.354 (60.735) | 727.130 (43.000) | 783.328 (46.155) | 880.822 (60.298)
Statistical Analysis 1: Comparison: Water Control vs 2g Capsules; Test type: Other; p = 0.0509, t-test, 2 sided
Statistical Analysis 2: Comparison: Water Control vs 4g Capsules; Test type: Other; p = 0.5016, t-test, 2 sided

8. Other Pre Specified Outcome: Effect of Axulin in Lean vs. Overweight Participants
Description: Percentage change in blood glucose area under the curve (AUC) in lean participants compared to overweight participants.
Time Frame: 0, 15, 30, 45, 60, 90, and 120 minutes post-dose
Population: Arms/Groups are provided as appropriate. The analysis of other outcome measures is based on all randomized subjects who received this intervention and for whom the outcome data is known. There is no missing value imputation.
Measure: Mean (Standard Error); unit: mmol x min/L
Groups:
- Water Control, Lean Participants: Lean Participants randomized to receive 250ml water.
- Water Control, Overweight Participants: Overweight Participants randomized to receive 250ml water.
- 2g Capsules, Lean Participants: Lean Participants randomized to receive 250ml water.with 8 x 250mg capsules containing Axulin powder plus 8 x 250mg placebo capsules.
- 2g Capsules, Overweight Participants: Overweight Participants randomized to receive 250ml water.with 8 x 250mg capsules containing Axulin powder plus 8 x 250mg placebo capsules.
- 4g Capsules, Lean Participants: Lean Participants randomized to receive 250ml water with 16 x 250mg capsules containing Axulin powder.
- 4g Capsules, Overweight Participants: Overweight Participants randomized to receive 250ml water with 16 x 250mg capsules containing Axulin powder.
- 2g Tablets, Lean Participants: Lean Participants randomized to receive 250ml water with 2 x 1g tablets containing Axulin powder.
- 2g Tablets, Overweight Participants: Overweight Participants randomized to receive 250ml water with 2 x 1g tablets containing Axulin powder.
- 4g Tablets, Lean Participants: Lean Participants randomized to receive 250ml water with 4 x 1g tablets containing Axulin powder.
- 4g Tablets, Overweight Participants: Overweight Participants randomized to receive 250ml water with 4 x 1g tablets containing Axulin powder.
- Placebo Capsules, Lean Participants: Lean Participants randomized to receive 250ml water.with 16 x 250mg placebo capsules.
- Placebo Capsules, Overweight Participants: Overweight Participants randomized to receive 250ml water.with 16 x 250mg placebo capsules.
Arm/Group | Water Control, Lean Participants | Water Control, Overweight Participants | 2g Capsules, Lean Participants | 2g Capsules, Overweight Participants | 4g Capsules, Lean Participants | 4g Capsules, Overweight Participants | 2g Tablets, Lean Participants | 2g Tablets, Overweight Participants | 4g Tablets, Lean Participants | 4g Tablets, Overweight Participants | Placebo Capsules, Lean Participants | Placebo Capsules, Overweight Participants
Number analyzed (Participants) | 9 | 11 | 9 | 11 | 9 | 11 | 9 | 11 | 9 | 11 | 9 | 11
mmol x min/L | 337.704 (26.343) | 264.474 (31.965) | 286.425 (30.944) | 230.891 (35.892) | 291.083 (50.563) | 206.168 (32.895) | 326.517 (34.054) | 324.941 (48.047) | 358.513 (38.841) | 253.858 (33.223) | 290.325 (54.912) | 243.699 (39.663)
Statistical Analysis 1: Comparison: 2g Capsules, Lean Participants vs 2g Capsules, Overweight Participants; Test type: Other; p = 0.8444, t-test, 2 sided
Statistical Analysis 2: Comparison: 4g Capsules, Lean Participants vs 4g Capsules, Overweight Participants; Test type: Other; p = 0.9681, t-test, 2 sided
Statistical Analysis 3: Comparison: 2g Tablets, Lean Participants vs 2g Tablets, Overweight Participants; Test type: Other; p = .1022, t-test, 2 sided
Statistical Analysis 4: Comparison: 4g Tablets, Lean Participants vs 4g Tablets, Overweight Participants; Test type: Other; p = .3738, t-test, 2 sided
Statistical Analysis 5: Comparison: Water Control, Lean Participants vs 2g Capsules, Lean Participants; Test type: Other; Mean Difference (Net) = -13.123, Standard Error of Mean 8.550 — Percentage Change from Control
Statistical Analysis 6: Comparison: Water Control, Overweight Participants vs 2g Capsules, Overweight Participants; Test type: Other; Mean Difference (Net) = -10.362, Standard Error of Mean 10.387 — Percentage Change from Control
Statistical Analysis 7: Comparison: Water Control, Lean Participants vs 4g Capsules, Lean Participants; Test type: Other; Mean Difference (Net) = -13.738, Standard Error of Mean 13.463 — Percentage Change from Control
Statistical Analysis 8: Comparison: Water Control, Overweight Participants vs 4g Capsules, Overweight Participants; Test type: Other; Mean Difference (Net) = -12.929, Standard Error of Mean 14.282 — Percentage Change from Control

9. Other Pre Specified Outcome: Effect of Capsules vs. Tablets
Description: Percentage change in blood glucose area under the curve (AUC) elicited by capsules compared to the same dose of tablets.
Time Frame: 0, 15, 30, 45, 60, 90, and 120 minutes post-dose
Population: The analysis of the outcome measure is based on all randomized participants who received this intervention and for whom the outcome data is known. There is no missing value imputation.
Measure: Mean (Standard Error); unit: mmol x min/L
Arm/Group | Water Control | 2g Capsules | 2g Tablets | 4g Capsules | 4g Tablets | Placebo Capsules
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
mmol x min/L | 297.428 (22.296) | 255.881 (24.383) | 325.650 (29.800) | 244.380 (29.859) | 300.953 (27.350) | 264.681 (32.481)
Statistical Analysis 1: Comparison: 2g Capsules vs 2g Tablets; Test type: Other; p = 0.0111, t-test, 2 sided
Statistical Analysis 2: Comparison: 4g Capsules vs 4g Tablets; Test type: Other; p = 0.1684, t-test, 2 sided
Statistical Analysis 3: Comparison: Water Control vs 2g Capsules; Test type: Other; Mean Difference (Net) = -11.604, Standard Error of Mean 6.722 — Percentage Change from Control
Statistical Analysis 4: Comparison: Water Control vs 2g Tablets; Test type: Other; Mean Difference (Net) = 12.755, Standard Error of Mean 8.489 — Percentage Change from Control
Statistical Analysis 5: Comparison: Water Control vs 4g Capsules; Test type: Other; Mean Difference (Net) = -13.293, Standard Error of Mean 9.664 — Percentage Change from Control
Statistical Analysis 6: Comparison: Water Control vs 4g Tablets; Test type: Other; Mean Difference (Net) = 2.526, Standard Error of Mean 5.813 — Percentage Change from Control

10. Post Hoc Outcome: Blood Glucose Change From Baseline in the Water Control Compared to the Placebo Capsules at 90 Minutes for All Participants
Description: Change from baseline (CFB) in blood glucose will be computed at 90 minutes. The CFB results for the water control and the placebo capsule treatments will be subjected to a paired t-test examining whether the mean difference between the two sets of observations is equal to zero.
Time Frame: From Baseline at 90 minutes
Population: The analysis of the outcome measure is based on all randomized participants who received this intervention and for whom the outcome data is known. The comparison is between the water control and the placebo capsules only. There is no missing value imputation.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Water Control | Placebo Capsules
Number analyzed (Participants) | 20 | 20
mmol/L | 2.475 (0.2736) | 1.953 (0.2969)
Statistical Analysis 1: Comparison: Water Control vs Placebo Capsules; Test type: Other; p = 0.0374, t-test, 2 sided; Percentage Change from Control = -21.09

11. Post Hoc Outcome: 60-Minute Blood Glucose Area Under the Curve (AUC)
Description: Incremental area under the blood glucose response curve (AUC) will be computed using the values recorded at 60 minutes and beyond. The blinded AUC results for the Axulin capsule treatments and the water control will be subjected to repeated measures analysis of variance (ANOVA) examining for the main effects of treatment and participant-group, and treatment*group interaction. After demonstration of significant heterogeneity among the 3 coded treatments, differences between individual means will be assessed using Tukey's test to adjust for multiple comparisons.
Time Frame: 1-2 hours post-dose
Population: The analysis of other outcome measures is based on all randomized subjects who received this intervention and for whom the outcome data is known. There is no missing value imputation.
Measure: Mean (Standard Error); unit: mmol x min/L
Arm/Group | Water Control | 2g Capsules | 4g Capsules | Placebo Capsules | 2g Tablets | 4g Tablets
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
mmol x min/L | 139.300 (13.533) | 105.566 (11.417) | 104.450 (15.392) | 118.316 (15.907) | 153.618 (18.640) | 135.475 (16.844)
Statistical Analysis 1: Comparison: Water Control vs 2g Capsules; Test type: Other; p = 0.0098, t-test, 2 sided; Percentage Change from Control = -24.22
Statistical Analysis 2: Comparison: Water Control vs 4g Capsules; Test type: Other; p = 0.0391, t-test, 2 sided; Percentage Change from Control = -25.02

12. Post Hoc Outcome: Blood Glucose Change From Baseline at 90 and 120 Minutes in All Participants
Description: Change from baseline (CFB) in blood glucose will be computed at 90 and 120 minutes. The CFB results for the capsule treatments and the water control will be subjected to a paired t-test examining whether the mean difference between the two sets of observations is equal to zero.
Time Frame: From Baseline at 90 and 120 minutes
Population: as for outcome 11
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Water Control | 2g Capsules | 4g Capsules | Placebo Capsules | 2g Tablets | 4g Tablets
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
mmol/L
  90-Minute Blood Glucose CFB | 2.475 (0.274) | 1.577 (0.252) | 1.653 (0.291) | 1.953 (.297) | 2.338 (.378) | 2.089 (.289)
  120-Minute Blood Glucose CFB | 1.469 (0.245) | 0.686 (0.249) | 0.790 (0.228) | 1.032 (.258) | 1.453 (.256) | 1.507 (.313)
Statistical Analysis 1: Comparison: Water Control vs 2g Capsules; Change from baseline (CFB) in blood glucose will be computed at 90 minutes. The CFB results for the capsule treatments and the water control will be subjected to a paired t-test examining whether the mean difference between the two sets of observations is equal to zero; Test type: Other; p = 0.0034, t-test, 2 sided; Percentage Change from Control = -36.28
Statistical Analysis 2: Comparison: Water Control vs 4g Capsules; [analysis description as in outcome 12, analysis 1]; Test type: Other; p = 0.0058, t-test, 2 sided; Percentage Change from Control = -33.21
Statistical Analysis 3: Comparison: Water Control vs 2g Capsules; Change from baseline (CFB) in blood glucose will be computed at 120 minutes. The CFB results for the capsule treatments and the water control will be subjected to a paired t-test examining whether the mean difference between the two sets of observations is equal to zero; Test type: Other; p = 0.0016, t-test, 2 sided; Percentage Change from Control = -53.27
Statistical Analysis 4: Comparison: Water Control vs 4g Capsules; [analysis description as in outcome 12, analysis 3]; Test type: Other; p = 0.0125, t-test, 2 sided; Percentage Change from Control = -46.19

13. Post Hoc Outcome: Blood Glucose Change From Baseline at 90 and 120 Minutes in Lean Participants
Description: Change from baseline (CFB) in blood glucose will be computed at 90 and 120 minutes for the Lean Participants. The CFB results for the capsule treatments and the water control will be subjected to a paired t-test examining whether the mean difference between the two sets of observations is equal to zero.
Time Frame: From Baseline at 90 and 120 minutes
Population: as for outcome 8
Measure: Mean (Standard Error); unit: mmol/L
Groups:
- Water Control: Lean Participants randomized to receive 250ml water.
- 2g Capsules: Lean Participants randomized to receive 250ml water.with 8 x 250mg capsules containing Axulin powder plus 8 x 250mg placebo capsules.
- 4g Capsules: Lean Participants randomized to receive 250ml water with 16 x 250mg capsules containing Axulin powder.
- Placebo Capsules: Lean Participants randomized to receive 250ml water.with 16 x 250mg placebo capsules.
- 2g Tablets: Lean Participants randomized to receive 250ml water with 2 x 1g tablets containing Axulin powder.
- 4g Tablets: Lean Participants randomized to receive 250ml water with 4 x 1g tablets containing Axulin powder.
Arm/Group | Water Control | 2g Capsules | 4g Capsules | Placebo Capsules | 2g Tablets | 4g Tablets
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
mmol/L
  90-Minute Blood Glucose CFB in Lean Participants | 2.902 (0.238) | 1.992 (0.379) | 2.022 (0.505) | 2.546 (.457) | 2.542 (.366) | 2.818 (.426)
  120-Minute Blood Glucose CFB in Lean Participants | 2.232 (0.206) | 1.340 (0.361) | 1.299 (0.366) | 1.710 (.438) | 1.857 (.359) | 2.479 (.354)
Statistical Analysis 1: Comparison: Water Control vs 2g Capsules; [analysis description as in outcome 12, analysis 1]; Test type: Other; p = 0.0788, t-test, 2 sided; Percentage Change from Control = -31.36
Statistical Analysis 2: Comparison: Water Control vs 4g Capsules; [analysis description as in outcome 12, analysis 1]; Test type: Other; p = 0.0887, t-test, 2 sided; Percentage Change from Control = -30.32
Statistical Analysis 3: Comparison: Water Control vs 2g Capsules; [analysis description as in outcome 12, analysis 3]; Test type: Other; p = 0.0266, t-test, 2 sided; Percentage Change from Control = -39.96
Statistical Analysis 4: Comparison: Water Control vs 4g Capsules; [analysis description as in outcome 12, analysis 3]; Test type: Other; p = 0.0455, t-test, 2 sided; Percentage Change from Control = -41.80

14. Post Hoc Outcome: Blood Glucose Change From Baseline at 90 and 120 Minutes in Overweight Participants
Description: Change from baseline (CFB) in blood glucose will be computed at 90 and 120 minutes for the Obese/Overweight Participants. The CFB results for the capsule treatments and the water control will be subjected to a paired t-test examining whether the mean difference between the two sets of observations is equal to zero.
Time Frame: From Baseline at 90 and 120 minutes
Population: as for outcome 8
Measure: Mean (Standard Error); unit: mmol/L
Groups:
- Water Control: Overweight Participants randomized to receive 250ml water.
- 2g Capsules: Overweight Participants randomized to receive 250ml water.with 8 x 250mg capsules containing Axulin powder plus 8 x 250mg placebo capsules.
- 4g Capsules: Overweight Participants randomized to receive 250ml water with 16 x 250mg capsules containing Axulin powder.
- Placebo Capsules: Overweight Participants randomized to receive 250ml water.with 16 x 250mg placebo capsules.
- 2g Tablets: Overweight Participants randomized to receive 250ml water with 2 x 1g tablets containing Axulin powder.
- 4g Tablets: Overweight Participants randomized to receive 250ml water with 4 x 1g tablets containing Axulin powder.
Arm/Group | Water Control | 2g Capsules | 4g Capsules | Placebo Capsules | 2g Tablets | 4g Tablets
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11
mmol/L
  90-Min Blood Glucose CFB, Overweight Participants | 2.126 (0.441) | 1.237 (0.316) | 1.351 (0.326) | 1.469 (.340) | 2.171 (.632) | 1.491 (.301)
  120-Min Blood Glucose CFB, Overweight Participants | 0.844 (0.305) | 0.151 (0.257) | 0.373 (0.230) | .477 (.190) | 1.122 (.342) | .711 (.338)
Statistical Analysis 1: Comparison: Water Control vs 2g Capsules; [analysis description as in outcome 12, analysis 1]; Test type: Other; p = 0.0261, t-test, 2 sided; Percentage Change from Control = -41.82
Statistical Analysis 2: Comparison: Water Control vs 4g Capsules; [analysis description as in outcome 12, analysis 1]; Test type: Other; p = 0.0391, t-test, 2 sided; Percentage Change from Control = -36.45
Statistical Analysis 3: Comparison: Water Control vs 2g Capsules; [analysis description as in outcome 12, analysis 3]; Test type: Other; p = 0.0372, t-test, 2 sided; Percentage Change from Control = -82.11
Statistical Analysis 4: Comparison: Water Control vs 4g Capsules; [analysis description as in outcome 12, analysis 3]; Test type: Other; p = 0.1631, t-test, 2 sided; Percentage Change from Control = -55.81

15. Post Hoc Outcome: Insulin Change From Baseline at 90 Minutes in All Participants
Description: Change from baseline (CFB) in insulin will be computed at 90 minutes. The CFB results for the capsule treatments and the water control will be subjected to a paired t-test examining whether the mean difference between the two sets of observations is equal to zero.
Time Frame: From Baseline at 90 minutes
Population: as for outcome 11
Measure: Mean (Standard Error); unit: uU/mL
Arm/Group | Water Control | 2g Capsules | 4g Capsules | Placebo Capsules | 2g Tablets | 4g Tablets
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
uU/mL | 48.345 (10.046) | 25.896 (4.174) | 38.851 (12.260) | 38.179 (6.175) | 37.152 (5.383) | 38.388 (7.536)
Statistical Analysis 1: Comparison: Water Control vs 2g Capsules; Change from baseline (CFB) in insulin will be computed at 90 minutes. The CFB results for the capsule treatments and the water control will be subjected to a paired t-test examining whether the mean difference between the two sets of observations is equal to zero; Test type: Other; p = 0.0303, t-test, 2 sided; Percentage Change from Control = -46.43
Statistical Analysis 2: Comparison: Water Control vs 4g Capsules; [analysis description as in outcome 15, analysis 1]; Test type: Other; p = 0.4283, t-test, 2 sided; Percentage Change from Control = -19.64

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each participant from the time informed consent was signed through study completion; April 26, 2017 - June 21, 2017, an average of 2 months.
Description: Serious classification based on the FDA regulatory definition of a serious Adverse Event.
Groups:
- Water Control, Lean Participants; Water Control, Overweight/Obese Participants: Participants randomized to receive 250ml water.
- Placebo Capsules, Lean Participants; Placebo Capsules, Overweight/Obese Participants: Participants randomized to receive 250ml water.with 16 x 250mg placebo capsules.
- 2g Capsules, Lean Participants; 2g Capsules, Overweight/Obese Participants: Participants randomized to receive 250ml water.with 8 x 250mg capsules containing Axulin powder plus 8 x 250mg placebo capsules.
- 4g Capsules, Lean Participants; 4g Capsules, Overweight/Obese Participants: Participants randomized to receive 250ml water with 16 x 250mg capsules containing Axulin powder.
- 2g Tablets, Lean Participants; 2g Tablets, Overweight/Obese Participants: Participants randomized to receive 250ml water with 2 x 1g tablets containing Axulin powder.
- 4g Tablets, Lean Participants; 4g Tablets, Overweight/Obese Participants: Participants randomized to receive 250ml water with 4 x 1g tablets containing Axulin powder.
Arm/Group | Water Control, Lean Participants | Water Control, Overweight/Obese Participants | Placebo Capsules, Lean Participants | Placebo Capsules, Overweight/Obese Participants | 2g Capsules, Lean Participants | 2g Capsules, Overweight/Obese Participants | 4g Capsules, Lean Participants | 4g Capsules, Overweight/Obese Participants | 2g Tablets, Lean Participants | 2g Tablets, Overweight/Obese Participants | 4g Tablets, Lean Participants | 4g Tablets, Overweight/Obese Participants
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11 | 0/9 | 0/11 | 0/9 | 0/11 | 0/9 | 0/11 | 0/9 | 0/11 | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 0/9 | 0/11 | 0/9 | 0/11 | 0/9 | 0/11 | 0/9 | 0/11 | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 0/9 | 0/11 | 0/9 | 0/11 | 0/9 | 0/11 | 0/9 | 0/11 | 0/9 | 0/11

LIMITATIONS AND CAVEATS:
Note: The dissolution time for the tablets is substantially longer (>60 min) than it is for the capsules, so it would not be expected that the tablet formulation would exhibit a pharmacologic response if administered only 40 minutes before the GTT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT03135015/Prot_SAP_000.pdf